CLINICAL TRIAL: NCT03722979
Title: Study of the Expression of Endoplasmic Reticulum Stress During Extracorporeal Circulation in Humans
Acronym: STRECH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017/179/HP
Record Dates: First submitted 2018-10-25; First posted 2018-10-29 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Cardiac Surgery
MeSH Terms: interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Other)
  Interventions: Procedure: Cardiac surgery

INTERVENTIONS:
Procedure: Cardiac surgery — The study will enroll patients having a planned cardiac surgery under extracorporeal circulation (CEC)

SUMMARY:
The links between systemic inflammation, endothelial dysfunction and endoplasmic reticulum (ER) stress in pre-clinical models make it an interesting potential therapeutic target, but there are no data describing SRE during severe inflammation in humans .

For an approach to the study of SRE in humans in a situation of systemic inflammation, the analysis of patients benefiting from an extra-corporeal circulation for a programmed cardiac surgery would allow a study under well described conditions of inflammation, standardized, with the possibility for each patient to be his own witness. Compared to a situation of secondary inflammation (sepsis, acute pancreatitis, trauma ...) the analysis of the patients under CEC allows more precise description of the kinetics of the activation of the SRE because the beginning of the inflammatory mechanism is known with precision.

ELIGIBILITY:
Inclusion Criteria:

* Major patient (age ≥ 18 years)
* Patient undergoing cardiac surgery under extracorporeal circulation (duration of planned CEC > 1h)
* Informed person, having read and signed his consent preoperatively no later than the day before the procedure.
* Person affiliated with a social security scheme
* Effective contraception in women of childbearing potential. For menopausal women, the diagnosis of menopause will be based on the gynecological history of the patient (age> 50 years + amenorrhea for more than 12 months).

Exclusion Criteria:

* Patient with urgent cardiac surgery
* Patient with cardiac surgery without extracorporeal circulation
* Patient with surgery under "mini-CEC"
* Patient with simple aortic valve replacement or single / double coronary artery bypass (CEC duration typically <1h)
* Patient with chronic autoimmune inflammatory disease, eg lupus, rheumatoid arthritis, inflammatory bowel disease ...
* Patient with progressive neoplastic disease
* Patient with underlying heart disease with left ventricular ejection fraction <30%
* Pregnant or lactating woman
* Person deprived of liberty by an administrative or judicial decision or protected major subject (under tutorship or curatorship)
* Patient participating in another interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-07-07 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-03-06 (Actual)

PRIMARY OUTCOMES:
Study of the variation of a marker of endoplasmic reticulum stress, between the pre- extracorporeal circulation (CEC) sample and the sample taken 2 hours after the release of extracorporeal circulation | 2 hours after the release of extracorporeal circulation
  ELISA technique (comparison of protein levels) + quantitative RT-PCR (comparison of normalized mRNA expression concentrations relative to a control gene).

CONTACTS AND LOCATIONS:
Locations (1):
- ROUEN Hospital University, Rouen, France